CLINICAL TRIAL: NCT01231035
Title: REsponsiveness to CLOpidogrel and Stent-related Events in Acute Coronary. Reclose 2-ACS Registry
Brief Title: REsponsiveness to CLOpidogrel and Stent-related Events in Acute Coronary Syndromes (RECLOSE 2 - ACS)
Acronym: RECLOSE2-ACS
Status: Completed | Type: Observational
Sponsor: Careggi Hospital (Other)
Responsible Party: David Antoniucci, Director of Invasive Cardiology Division, Careggi Hospital
Other Study IDs: RECLOSE 2-ACS; Apice (Other Grant/Funding Number: Ministry of Health, Italy)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Acute Cardiac Syndrome; Stent Thrombosis; Platelet Function; Antiplatelet Therapy
Keywords: acute cardiac syndrome; stent thrombosis; platelet function; antiplatelet therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of the project is to assess the long-term prognostic impact of residual platelet reactivity after optimal antiplatelet therapy in a large cohort of patients with acute coronary syndrome undergoing invasive strategy.

Follow-up length will be at least 24 months. The primary end-point of the study will be a composite of death, myocardial infarction, urgent target vessel revascularization, stent thrombosis or stroke.

DETAILED DESCRIPTION:
This study is mainly based on a registry of 2000 consecutive patients with acute coronary syndrome who received invasive treatment and for whom platelet reactivity after clopidogrel treatment will be prospectively assessed.

In the acute phase, blood samples for platelet reactivity assessment will be obtained 12 to 18 hours from 600 mg clopidogrel loading. Platelet-rich plasma, obtained by centrifuging whole blood for 10 min at 200 g, was stimulated with 10 M adenosine 5'-diphosphate (ADP) and residual aggregation will be assessed using a APACT 4 light transmittance aggregometer. Platelet aggregation (according to the Born's method) will be evaluated considering the maximal percentage of platelet aggregation in response to stimulus. Patients with platelet aggregation by 10 µmol ADP ≥ 90th percentile of controls (70%) will be defined as non-responders. The assessment of platelet reactivity will be repeated at 6 months. The importance of concomitant aspirin resistance will be also evaluated in such of patients.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome
* invasive treatment

Exclusion Criteria:

* in-hospital death that was not due to stent thrombosis,
* anticipated poor compliance to dual antipletelet treatment for at least 6 months,
* premature discontinuation of clopidogrel therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute coronary syndrome who received invasive treatment and for whom platelet reactivity after clopidogrel treatment will be prospectively assessed.
Sampling Method: Probability Sample
Enrollment: 1789 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
long-term prognostic impact of residual platelet reactivity | 24 months
  to assess the long-term prognostic impact of residual platelet reactivity after optimal antiplatelet therapy in a large cohort of patients with acute coronary syndrome undergoing invasive strategy.

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Study Director — Careggi Hospital, Division of Invasive Cardiology
Locations (1):
- Careggi Hospital, Department of Heart and Vessels, Florence, Italy

REFERENCES:
- [Background] Parodi G, Marcucci R, Valenti R, Gori AM, Migliorini A, Giusti B, Buonamici P, Gensini GF, Abbate R, Antoniucci D. High residual platelet reactivity after clopidogrel loading and long-term cardiovascular events among patients with acute coronary syndromes undergoing PCI. JAMA. 2011 Sep 21;306(11):1215-23. doi: 10.1001/jama.2011.1332. PMID 21934054